CLINICAL TRIAL: NCT00970333
Title: Evaluation of [18F] FEPPA and PET as a Marker of Inflammation in Subjects With Neurological Conditions
Brief Title: Evaluation of [18F] FEPPA and PET Imaging as a Marker of Inflammation in Subjects With Neurological Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FEPPA 001
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Alzheimer Disease; Parkinson Disease; Multiple Sclerosis
Keywords: Alzheimer disease; Parkinson disease; Multiple Sclerosis
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Multiple Sclerosis | interventions — N-(2-((N-(4-phenoxypyridin-3-yl)acetamido)methyl)phenoxy)ethyl fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- assess [18F]-FEPPA PET imaging (Experimental)
  Interventions: Drug: [18F]-FEPPA

INTERVENTIONS:
Drug: [18F]-FEPPA — Subjects will be injected with up to 5 mCi and not to exceed 5.5mCi (not >10% of 5 mCi limit) of [18F]-FEPPA followed by serial PET imaging

SUMMARY:
Ultimately a marker of microglial activation could be used for large-scale quantitative brain imaging trials in Alzheimer Disease (AD), Parkinson Disease (PD) or Multiple Sclerosis (MS), specifically to investigate the agent as an objective biomarker in treatments aimed at reducing inflammatory changes in these conditions. The significance of this work lies in applying state-of-art quantitative neuroimaging tools to develop a relevant biomarker in individuals with neurodegenerative diseases with the intention of using this efficiently in large clinical imaging trials.

DETAILED DESCRIPTION:
The adaptation of imaging agents like [18F]-FEPPA as a biomarker of microglial activation in neurodegenerative and neuroinflammatory diseases requires human validation studies. Expanding upon our previous work with B-amyloid ligands (123I-IMPY, 123I MNI-187) for AD and dopamine transporter ligands (123I B-CIT, Altropane) for PD, we desire to develop and characterize [18F]-FEPPA as a potential marker for microglial activation in association with neuronal damage that may be applicable to multiple neurodegenerative and inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease patients will be recruited for this study. The following criteria will be met for inclusion of AD subjects in this study:

  * The participant is 50 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of probable Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
  * Clinical Dementia Rating Scale score ≤ 2.
  * Modified Hachinski Ischemia Scale score of ≤ 4.
  * For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-FEPPA injection.

Exclusion Criteria:

* Alzheimer's subjects will be excluded from participation for the following reasons:

  * The subject has a history of significant cerebrovascular disease.
  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy

Inclusion Criteria:

* The following criteria will be met for inclusion of PD subjects in this study:

  * The participant is 30 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of Parkinson disease (at least two of the three cardinal symptoms: resting tremor, rigidity, bradykinesia).
  * Hoehn and Yahr ≤4.
  * For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-FEPPA injection.

Exclusion Criteria:

* Parkinson's subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy

Inclusion Criteria:

* Multiple Sclerosis Subject Selection. Subjects who have a clinical diagnosis of Multiple Sclerosis (MS) will be recruited for this study. The following criteria will be met for inclusion of MS subjects in this study:

  * The participant is 18 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of Multiple Sclerosis (per the 2005 Revised McDonald Criteria; Polman, et al., 2005).
  * Kurtzke Expanded Disability Status Scale (EDSS) ≤ 7.5.
  * For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-FEPPA injection.

Exclusion Criteria:

* MS subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, [18F]-FEPPA. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Instiute for Neurodegenerative Disorders, New Haven, Connecticut, United States